CLINICAL TRIAL: NCT05254444
Title: Samaki Salama: Securing Small-scale Fisheries in Kenya for Healthy Nutrition and Ecosystems
Brief Title: Samaki Salama: Small-scale Fisheries for Healthy Nutrition and Ecosystems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Rhode Island (Other); Pwani University (Unknown); Egerton University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 7200AA18CA00030
Record Dates: First submitted 2021-06-15; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Malnutrition, Child; Growth; Stunting, Nutritional
Keywords: Social marketing; Fish; Animal source food; Complementary feeding; Sustainable fishing
MeSH Terms: conditions — Child Nutrition Disorders; Growth Disorders | interventions — Social Marketing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Control (No Intervention): No activities will take place in group 1.
- Group 2: Social Marketing (Experimental): Households in this arm will receive a multi-tiered social marketing campaign focusing on sustainable fish nutrition, dietary diversity and food safety.
  Interventions: Behavioral: Social marketing
- Group 3: Social Marketing + Gear Modification (Experimental): Households in this arm will receive a bundled intervention of the social marketing campaign as well as modified fishing gear (basket traps with fish escape gaps) and training on proper utilization and management.
  Interventions: Behavioral: social marketing + gear modification

INTERVENTIONS:
Behavioral: Social marketing — Multi-tiered nutrition social marketing intervention focused on sustainable fish nutrition, dietary diversity and food safety.
  Arms: Group 2: Social Marketing
Behavioral: social marketing + gear modification — Multi-tiered nutrition social marketing intervention plus fishing gear modification (basket trap) and training.
  Arms: Group 3: Social Marketing + Gear Modification

SUMMARY:
The purpose of this study is to test the effectiveness of a bundled intervention to address malnutrition and its intersections with nutrition security and fisheries sustainability in Kilifi, Kenya.

DETAILED DESCRIPTION:
One in five young children globally suffer the consequences of stunted growth and development, while millions experience deficiencies in zinc, iron, iodine, vitamins A and B12, nutrients found bioavailable in fish foods. Small-scale fisheries (SSF) have the potential to generate wealth and augment fish consumption while being environmentally sustainable if appropriate systems are in place. However, those engaged in SSF are often marginalized by large industrial fisheries and other factors. Coastal communities in Kenya are dominated by SSF and are among the poorest and most malnourished globally. To address these critical issues, investigators aim to test the effectiveness of a bundled intervention to address malnutrition and its intersections with nutrition security and fisheries sustainability.

A matched intervention/control study will be conducted to examine the multifaceted Samaki Salama ("fish security" in Kiswahili) intervention in Kilifi, Kenya. The matched communities will be divided into three groups: (1) control; (2) multi-tiered nutrition social marketing intervention to fishers, mothers, and health workers; (3) multi-tiered nutrition social marketing intervention plus fisher gear modification and training.

A total of 8 communities will be matched based on based on location (rural), livelihoods and child nutritional status into control (n=4) and intervention (n=4) groups. Participants from 400 small-scale fisher households will be recruited and enrolled by Kenyan partners from Egerton University and Pwani University using the eligibility criteria. Group 1 (n=200 households) will be the control group. Group 2 (n=100 households) will receive a multi-tiered nutrition social marketing intervention focused on promoting dietary diversity and fish food consumption specifically among infants, young children and women of reproductive age. The nutrition intervention will target fishers, mother and health workers and involve monthly communications of key nutrition messages across a range of platforms including mobile phone messaging through WhatsApp or SMS, social media, radio, t-shirts, stickers, flyers, cooking classes, meetings of mother's groups and other convening opportunities. Group 3 (n=100 households) will receive a bundled intervention of the multi-tiered nutrition social marketing intervention plus fisher gear modification and training. Fishers from Group 3 will receive modified fishing gear (traps) designed specifically to improve harvest efficiency and promote sustainable fish populations. Training on modified gear use will be administered through local fishing cooperatives.

Investigators hypothesize that the combined impact of the targeted social marketing and fisher trap interventions will improve the diet, health and nutritional status of children as well increase fisheries yield and fisher's earnings in intervention communities. Specific hypotheses of primary and secondary outcomes are as follows:

Hypotheses: primary outcomes

* The children in the intervention groups (combined groups 2 and 3) with have increased height-for-age Z score (HAZ) by 0.20 compared to children in the control (group 1).
* The children in the intervention groups (combined groups 2 and 3) with have increased weight-for-age Z score (WAZ) by 0.10 compared to children in the control (group 1).
* The children in the intervention groups (combined groups 2 and 3) with have increased fish food intakes by 100 g compared to children in the control (group 1).
* Fishers in the group 3 will have significantly increased fisheries yields of mature fish compared to fishers in the control (group 1).

Hypotheses: secondary outcomes

* The children in the intervention groups (combined 2 and 3) with have increased dietary diversity by 1.2 compared to children in the control (group 1).
* The children in the intervention groups (combined 2 and 3) with have reduced diarrheal morbidity by 5 percentage points compared to children in the control (group 1).
* Fishers in group 3 will have significantly increased earnings compared to fishers in the control (group 1).

ELIGIBILITY:
Inclusion Criteria:

* A household member works in small-scale fisheries (self-employed fishers)
* At least one child in the household aged 6-60 months
* At least one member of the household owns a mobile phone
* Provision of signed and dated informed consent form
* For children, informed assent and parental informed consent to participate in the study
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* No household member works in small-scale fisheries (self-employed fishers)
* No child in the household aged 6-60 months
* No members of the household own a mobile phone
* Declines to sign the informed consent
* Index child is severely malnourished
* Lives outside the study area
* Participation in another nutrition or fisheries intervention study within April 2021 - June 2022

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change in child weight | Change from baseline weight-for-age (WAZ) at 12 months
  Child weight in kilograms. A weight-for-age Z score (WAZ), a measure of underweight, will be calculated using weight and date of birth.
Change in child height | Change from baseline height-for-age (HAZ) at 12 months
  Child height in centimeters. A height-for-age Z score (HAZ), a measure of stunting, using height and date of birth
Change in child fish foods intake | Change from baseline fish foods intake at 12 months
  Intake of fish foods assessed for children 6-60 months using a Kenya-specific semi-quantitative food frequency questionnaire (FFQ) that includes both 24-hour and 7-day recalls.
Change in fisheries yield | Change from baseline fisheries yield at 12 months
  Fisher's catch will be counted and weighed and identified at landing sites. Lengths of fish will be measured for a sub-sample of individuals (n=20). Monthly catch per unit effort (i.e. yield) will be calculated as the mean daily catch multiplied by the fishing days per month. Sustainable yields will be determined by comparing the initial yields versus the rate of change of yields for each landing site or Beach Management Unit (BMU).

SECONDARY OUTCOMES:
Child Dietary Diversity | Baseline and months 6 and 12
  Dietary intakes will be measured using Kenya-specific semi-quantitative food frequency questionnaire (FFQ). A comprehensive list of foods consumed in Kenya, and specifically along the coast, will be compiled along with ingredients in common dishes. This will be integrated into the survey as an FFQ for 24-hr intakes of youth and children ages 6-60 months. Findings from the FFQ will later be converted to the Feed the Future (FTF) indicators of minimum dietary diversity. Finally, infant and young child feeding practices (IYCF) practices will be assessed in accordance with the FTF minimum acceptable diet indicator.
Child Diarrheal Morbidity | Baseline and months 6 and 12
  Measured using mothers' reporting of acute diarrhea (3 or more liquid or semi-liquid stools in a 24-hour period over the last two weeks).
Fisheries Earnings | Baseline, regular intervals (5-10 times per month) for 12 months
  Data on fisher operational costs and revenue generation will be collected using surveys. Questions will be informed by cultural norms and objects such as food and equipment used as currency when Kenyan Shillings cannot be estimated (e.g. bags of rice).

CONTACTS AND LOCATIONS:
Overall Officials: Lora Iannotti, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Pwani University, Kilifi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be analyzed and stored on the REDCap platform and on Box, a secure, HIPAA and FERPA compliant data storage and sharing online platform. After the study is completed, the de-identified, archived data will be transmitted to the USAID Feed the Future Fish Innovation Lab for use by other researchers including those outside of the study.
  Data from this study may be requested from other researchers 2 years after the completion of the primary endpoint by contacting the PI from the sponsor University.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 years from the completion of primary endpoints.
Access Criteria: Researchers wanting to use the data would have to contact the PIs and explain their purpose for using the data.

REFERENCES:
- [Derived] Blackmore I, Wamukota A, Kamau-Mbuthia E, Humphries A, Lesorogol C, Cohn R, Sarange C, Mbogholi F, Obata C, Cheupe C, Cheupe J, Sherburne L, Chapnick M, Cartmill MK, Iannotti LL. Samaki Salama - Promoting healthy child growth and sustainable fisheries in coastal Kenya: A study protocol. Front Public Health. 2022 Oct 21;10:934806. doi: 10.3389/fpubh.2022.934806. eCollection 2022. PMID 36339158